CLINICAL TRIAL: NCT00114608
Title: Venous Blood Flow Velocity: Electrical Foot Stimulation Compared to Intermittent Pneumatic Compression of the Foot
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University at Buffalo (Other)
Responsible Party: Robert E. Kaplan, MD, Associate Clinical Professor, University at Buffalo School of Medicine and Biomedical Sciences
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY # 2
Record Dates: First submitted 2005-06-15; First posted 2005-06-16 (Estimated); Last update posted 2008-03-11 (Estimated); Status verified 2008-03

CONDITIONS: Deep Vein Thrombosis; Pulmonary Embolism
Keywords: Electrical foot stimulation; Intermittent pneumatic compression; Venous thromboembolism; Immobilization; Total hip replacement; Prolonged travel; Venous thromboembolic disease (VTE); Deep vein thrombosis (DVT); Pulmonary embolism (PE)
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism; Venous Thromboembolism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Electrical foot stimulation
  Interventions: Device: The Focus™ Neuromuscular Stimulation System

INTERVENTIONS:
Device: The Focus™ Neuromuscular Stimulation System — Electrical foot stimulation was produced by surface electrodes placed on the sole of the foot over the plantar muscle group. Electrical stimulation was delivered by The Focus™ Neuromuscular Stimulation System, Empi, Inc. (St. Paul, MN.) The crucial stimulus parameters were: biphasic symmetrical square wave at 50 pulses per second, phase duration of 300 microseconds, a starting ramp up time of 2 seconds and a finishing ramp down time of 2 seconds per stimulation cycle, and a stimulation cycle of 12 seconds "on" and 48 seconds "off" per minute. Stimulation was increased to an intensity just sufficient to create a slight visible muscle twitch. This level of intensity caused no evident discomfort in any of the subjects in our first study. Subjects were continually monitored throughout this study for any indication of discomfort.The Focus™ Neuromuscular Stimulation System created electrical stimulation of the plantar foot muscles.

SUMMARY:
Electrical stimulation of the foot can increase blood flow out of the leg. This increased blood flow can prevent blood clots from forming in the leg veins.

Blood clots in the leg veins can break off and form life-threatening blood clots in the lungs.

Intermittent external pneumatic (air) compression of the foot is already used to increase blood flow in at risk patients.

Hypothesis: Electrical stimulation of the foot increases blood flow out of the legs to the same degree as intermittent external pneumatic (air) compression of the foot.

DETAILED DESCRIPTION:
ABSTRACT Background: Venous stasis caused by immobility is an important risk factor for venous thromboembolic disease. This is especially true for orthopedic patients with multiple trauma and those undergoing other orthopedic procedures. A safe and convenient method for reducing venous stasis would be useful for preventing venous thrombosis in patients while in hospital and particularly after discharge during rehabilitation. In a prior study, we demonstrated that electrical stimulation of the foot was a safe and convenient method for counteracting venous stasis. In this study, we compare the effects on venous blood flow of intermittent pneumatic compression, an established method, to electrical stimulation of the foot.

Methods: 40 healthy volunteers aged 50 - 80 were seated for 4 hours during which they received mild electrical stimulation of the sole of the foot (plantar plexus of muscles) or intermittent pneumatic compression. Popliteal and femoral venous blood flow velocities were measured via Doppler ultrasound. Blood flow in the non-stimulated or non-compressed lower extremity served as a simultaneous control. Subjects completed a questionnaire regarding their acceptance and tolerance of both treatments.

INTRODUCTION Venous thrombosis and pulmonary embolism or venous thromboembolism (VTE) are important complications of medical and surgical conditions that are associated with prolonged immobilization. This is especially true for orthopedic patients with multiple trauma and those undergoing other orthopedic procedures. Immobilization is also a major contributor to the increased risk of VTE associated with prolonged air travel.

Despite good evidence that prophylaxis is effective, there is widespread under utilization of prophylaxis for VTE following major surgical procedures as well as medical conditions that produce weakness or prolonged bed rest. There is also good evidence that the risk of VTE continues for weeks after major orthopedic as well as other types of surgery. It is now recognized that VTE occurring in the hospital and outside the hospital setting is a single entity and that extended prophylaxis with anticoagulants reduces the risk.

Anticoagulant prophylaxis after hospital discharge although indicated in certain high risk groups is inconvenient since the recommended methods, LMWH and fondaparinux must be administered by subcutaneous injection and warfarin requires laboratory monitoring.

Physical methods that increase blood flow in the leg veins are effective for reducing venous thrombosis in high-risk hospitalized medical and surgical patients. These methods include: high intensity electrical calf stimulation during surgery, graduated compression stockings and intermittent pneumatic compression of the leg or foot. Of these, only graduated compression stockings, which are not very effective, can be used after hospital discharge. Graduated compression stockings, however, cannot be adapted to fit all leg shapes, may be improperly applied, have a tendency to slip down the leg and are found to be uncomfortable by many patients. High intensity electrical calf muscle stimulation is painful and can only be used during general anesthesia. AC powered external pneumatic compression can only be used while the patient is fully immobilized. Thus, alternative convenient methods are needed which can be used both in the immobilized and partly mobile patient, particularly after hospital discharge.

We have attempted to overcome the limitations of currently available physical devices by using mild electrical stimulation of the plantar muscles of the feet. Each electrical discharge elicits a foot twitch that causes the intrinsic foot muscles to contract. This contraction compresses the plantar plexus of veins, thereby increasing venous velocity in the popliteal and femoral veins that is transmitted proximally up the leg veins.

Our plantar foot stimulation device is powered by a 9-volt battery and small enough to be inserted into a sock. It has the potential to be worn while a patient is immobile, standing or walking, and therefore is suitable for use both during the initial period of immobilization and throughout convalescence.

In an earlier study we reported that mild electrical stimulation of the plantar foot muscles caused an increase in blood flow comparable to that produced by direct calf stimulation.

The aim of this new study is to determine if, over a 4 hour period, mild electrical stimulation of the plantar foot muscles increases venous blood flow velocity to the same degree as intermittent pneumatic compression (IPC) of the leg in both obese and non-obese subjects.

MATERIALS AND METHODS IRB approval and informed consent was obtained from all subjects. Forty healthy subjects (N = 40) between the ages of 50 to 80 participated in the study. Half of the subjects (N = 20) were non-obese with a Body Mass Index (BMI) < 30. The other half of the subjects (N = 20) were obese with a BMI > 30. Exclusion criterion included a prior history of deep vein thrombosis or pulmonary embolism, or any trauma or surgery involving any part of the lower extremities.

Subjects were studied over 2 sessions. At each session, subjects received either electrical foot stimulation or intermittent pneumatic compression of one foot. The other lower extremity served as a control. Subjects received either therapy at one session and the other therapy at a second session at least 48 hours later. The right or left leg of each subject was randomly assigned as the same control leg for both studies. The type of therapy given at the first session was also randomly assigned.

The study otherwise followed the protocol used in our initial study of electrical foot stimulation. Subjects were seated for 4 hours in chairs placed at a fixed distance apart. They were constantly monitored throughout the study to ensure that they remained seated. Subjects were allowed to use a bathroom located several feet away only twice during the 4 hour period. During the 4 hour study period subjects were offered a maximum of 16 ounces of fluid and a normal lunch.

Electrical foot stimulation was produced by surface electrodes placed on the sole of the foot over the plantar muscle group. Electrical stimulation was delivered by the Focus™ Neuromuscular Stimulation System, Empi, Inc. (St. Paul, MN.) The crucial stimulus parameters were: biphasic symmetrical square wave at 50 pulses per second, phase duration of 300 microseconds, a starting ramp up time of 2 seconds and a finishing ramp down time of 2 seconds per stimulation cycle, and a stimulation cycle of 12 seconds "on" and 48 seconds "off" per minute. Stimulation was increased to an intensity just sufficient to create a slight visible muscle twitch. This level of intensity caused no evident discomfort in any of the subjects in our first study. Subjects were continually monitored throughout this study for any indication of discomfort.

Intermittent pneumatic compression of the leg consisted of external intermittent pneumatic compression with a knee high device. A Tyco Healthcare Kendall Novamedix A-V impulse system® Model 6060 (Mansfield, MA 02048) was used. Operating parameters were: 130mmHg impulse pressure with a 3 second impulse duration; "Program Preset 1" for deep vein thrombosis prophylaxis. The compression followed the approved standard patient protocol used at our institution detailed in "Utilization of Intermittent Pneumatic Compression (IPC) Stockings for DVT Prophylaxis".

Popliteal and femoral venous peak blood flow velocities were measured bilaterally using a Doppler ultrasound device at 0, 15, 120, and 240 minutes. The same ultrasound technician obtained all Doppler studies on all subjects throughout the study. All Doppler tracings were be read by the same independent reader in a blinded fashion. Immediately following completion of each 4 hour session of electrical foot stimulation or intermittent pneumatic compression, subjects were asked to complete a brief questionnaire regarding their acceptance and tolerance of electrical stimulation or intermittent pneumatic compression.

STATISTICAL METHODS This study utilized a repeated measures design with two within group factors: time to measurement, and stimulation (stimulation, control). Stimulation groups [electrical foot stimulation and intermittent pneumatic compression (IPC)] were not independent. Blood flow measurements (at time = 120, 240) were analyzed with t tests and a mixed model. Within the mixed model, the group effect is a fixed effect, and the subject parameter is a random effect. The primary research question was the non-inferiority of the experimental treatment (electrical foot stimulation) relative to standard treatment (intermittent pneumatic compression). The non-inferiority index was 5.0 cm/sec; this index was formulated prior to analysis. The questionnaire results were analyzed using Fisher's Exact test. P-values that were less than 0.05 were considered to be statistically significant. All analyses were done with SAS 9.1, Cary, NC.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers

Exclusion Criteria:

* Venous or arterial disease of the lower limbs
* Cardiac pacemaker
* Known allergy to materials of surface electrodes
* Neurologic disorder
* Lower extremity fracture history
* History of joint replacement surgery
* Anticoagulation therapy other than aspirin

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-06; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Doppler venous blood flow velocity changes over 4 hours | Two, 4 hour sessions

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Kaplan, MD, Principal Investigator — University at Buffalo School of Medicine and Biomedical Sciences; James J Czyrny, MD, Principal Investigator — University at Buffalo School of Medicine and Biomedical Sciences
Locations (1):
- Erie County Medical Center, Buffalo, New York, United States

REFERENCES:
- [Background] Kaplan RE, Czyrny JJ, Fung TS, Unsworth JD, Hirsh J. Electrical foot stimulation and implications for the prevention of venous thromboembolic disease. Thromb Haemost. 2002 Aug;88(2):200-4. PMID 12195689